CLINICAL TRIAL: NCT05365815
Title: Black Midwives for Black Women: Maternity Care to Improve Trust and Attenuate Structural Racism
Brief Title: Melanated Group Midwifery Care (MGMC)
Acronym: MGMC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, Kylea Laina Liese, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CHAIRb 21120101; AD-2020C3-21229 (Other Grant/Funding Number: PCORI Foundation)
Record Dates: First submitted 2022-04-26; First posted 2022-05-09 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy Complications; Maternal Care Patterns; Patient Engagement
MeSH Terms: conditions — Pregnancy Complications; Patient Participation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The research team working on the effectiveness evaluation of group care is blinded to study condition and is charged with collecting the Aim 1 effectiveness data from the individuals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MGMC Intervention Group (Experimental): In the MGMC (intervention) group, pregnant women will participate in group prenatal care and have ~2-hour visits with the same two co-facilitators, a Black midwife and a Black care coordinator, along with 8-12 other Black women at a similar stage of pregnancy, for all prenatal and one postnatal care visits.
  The care coordinator will proactively engage with women throughout pregnancy and up to 12 months postpartum. The care coordinator helps women make appointments, sends reminders, and follows-up to ensure care was received, understood, and was appropriate. In the 3rd trimester, women in MGMC will be introduced to a community-based postpartum doula. The doula will make home visits once before birth and within the first 2 weeks postpartum; they will have approximately 50 contact hours available for 12 months postpartum for primarily in-person support, but they will be available by phone and text.
  Interventions: Behavioral: Melanated Group Midwifery Care
- Usual Care (No Intervention): In the usual care (comparator) group, pregnant women attend individually scheduled visits with a midwife or obstetrician for a physical assessment and counseling. Although this can vary by provider, continuity of care is rare and racial concordance is not a consideration. Referrals for medical or social services are given to the patient to complete in both prenatal and postnatal care.

INTERVENTIONS:
Behavioral: Melanated Group Midwifery Care — Racially concordant maternity care Group prenatal care Racially concordant nursing care coordination Postpartum doula support
  Arms: MGMC Intervention Group

SUMMARY:
This study is being conducted to determine if a multi-level intervention for delivering maternity care can improve patient trust and engagement among Black birthing people.

DETAILED DESCRIPTION:
Low-risk pregnant participants will be randomized into Melanated Group Midwifery Care or usual individualized obstetric care. In Melanated Group Midwifery Care (MGMC), Black women will receive prenatal care from a Black midwife in groups with the same 8-10 other Black women throughout pregnancy. In pregnancy and into the first year postpartum, MGMC patients will stay connected to the health system through a proactive care coordinator, who is a Black licensed nurse. For the first year after giving birth, patients in MGMC will also be supported by a trained postpartum doula.

All participants (intervention and usual care groups) will complete study measures that include validated surveys on patient trust, respect and engagement at 6 time points:

* 3 time points in pregnancy [baseline (<20 weeks), 26-28 weeks, and 35- 37 weeks] and
* 3 in the postpartum at 2-, 6-, and 12-months
* Additional qualitative interviews will be done to track the care received by medically and socially complex patients, including all who experience a severe maternal morbidity.

The investigators will also document how MGMC gets embedded in practice through a qualitative process evaluation.

ELIGIBILITY:
Inclusion criteria for patients:

* pregnant women who self-identify as Black on a standard prenatal intake form
* less than 20 weeks pregnant
* 15 years old or older
* present to the general obstetrics group at the University of Chicago Medical Center for their new prenatal visit
* speak and understand English

Inclusion criteria for providers:

• All black midwives, care coordinators, and community postpartum doulas at the University of Chicago are eligible to participate.

Exclusion criteria for patients:

* having a condition for which they present to a higher level of obstetrics care (e.g., maternal fetal medicine) for their new prenatal visit
* having a cognitive issue that impairs their ability to give informed consent.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 432 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Patient Engagement-Prenatal Adequacy | Birth (T3)
  Appropriate number (yes/no) and timing of prenatal visits (yes/no) documented in electronic medical records
Patient Engagement-Prenatal Adherence | Birth (T3)
  Five tests completed during prenatal period (yes/no), documented in electronic medical record
Patient Engagement-Postnatal adequacy | 1 year postpartum (T6)
  Appropriate number (yes/no) and timing of postnatal visits (yes/no) documented in electronic medical record

SECONDARY OUTCOMES:
Patient activation | Change from baseline through 12 months postpartum (T6)
  Patient Activation Measure (PAM), 13-item scale, range 0-100, Likert disagree strongly to agree strongly and not applicable. Assesses degree to which individuals take an active role in managing health and health care. Higher scores are more likely to understand that their active involvement is critical to their state of health and considered more ''in charge.'' The PAM has strong psychometric properties and is predictive of a wide range of health-related behaviors. Hibbard et al. report that a 4-point difference in PAM scores can be viewed as clinically significant.
Patient Autonomy | Change from baseline through 12 months postpartum (T6)
  Mothers Autonomy in Decision-Making Scale. 7 item scale, Likert completely disagree to completely agree. Assesses the degree to which patients were given decision-making for healthcare decisions, and if patients felt respected by providers. Higher scores indicate that providers supported patient autonomy and patient decision-making.
Provider Trust | Change from baseline through 12 months postpartum (T6)
  Trust in Physician Scale, 11 items, range 11-55, Likert 1-5; α =0.85-0.90.
Patient Satisfaction | Change from late pregnancy (35-37 gestational weeks) (T3) and 2 months postpartum (T4)
  22 items; 5-point Likert (excellent to poor); α =0.95. Excellent reliability and construct validity, taps six established dimensions of satisfaction (art of care, technical quality, access, physical environment, availability, and efficacy)
Mental Well Being | Change from baseline through 12 months postpartum (T6)
  Computerized Adaptive Testing - Mental Health: assessing depression, anxiety, suicidality, substance use disorder, and social determinants of health.
Respectful Care | Change from late pregnancy (35-37 gestational weeks) (T3) and 2 months postpartum (T4)
  Mothers on Respect index (MORi) quantifies women's sense of disrespect and dismissal when engaging in conversation with providers, 14 items, Likert, ranging from 1-strongly disagree to 6-strongly agree. α =0.94

OTHER OUTCOMES:
Medical Referrals | 12 months postpartum (T6)
  Referrals to higher acuity medical or obstetric care
Social Referrals | 12 months postpartum (T^)
  Referrals to higher acuity mental health or social services

CONTACTS AND LOCATIONS:
Overall Officials: Stacie L Geller, PhD, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No